CLINICAL TRIAL: NCT02686606
Title: A Randomised Controlled Crossover Trial to Investigate the Effect of Different Oral Nutritional Supplements on Fluid and Sodium Status in Patients With Short Bowel Intestinal Failure
Brief Title: A Trial to Investigate the Effect of Different Supplements on Fluid and Sodium Status in Short Bowel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NWLondonH
Record Dates: First submitted 2016-02-05; First posted 2016-02-19 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2021-03

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Ensure Plus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vital 1.5 (Experimental): 200ml orally over 30 minutes
  Interventions: Dietary Supplement: Vital 1.5
- Ensure Plus (Active Comparator): 200ml orally over 30 minutes
  Interventions: Dietary Supplement: Ensure Plus

INTERVENTIONS:
Dietary Supplement: Vital 1.5 — Oral nutritional supplement
  Arms: Vital 1.5
Dietary Supplement: Ensure Plus — Oral nutritional supplement
  Arms: Ensure Plus

SUMMARY:
Patients with short bowel intestinal failure are recommended to aim for a diet high in energy and protein. Some patients have difficulties in achieving recommended intakes and additional nutrition may be provided by oral nutritional supplements. There is very little research completed on which is the best oral nutritional supplement for patients. The aim of the study is to see the effect different oral nutritional supplements have on your stoma or fistula output and levels of hydration.

DETAILED DESCRIPTION:
After written consent is obtained, patients will be asked to fast from 12.00am on day one. At 08.00am patients will be asked to pass urine and to empty their stoma bag. After this they will be asked to drink 200ml of the ONS which they have been randomised to test on day one over a 30 minute period. Urine and intestinal output will be collected into two separate containers over the next 6 hours. During this time the patient will not be permitted to eat or drink other fluids. After 6 hours the patient will be able to eat and drink normally. The urine and intestinal output will be weighed and then an aliquot will be stored in a -20oC freezer before being sent for analysis. Day two is a washout day when the patient will be able to eat and drink normally. Day three will be the same as day one but the patient will have the other ONS that they did not have on day one. No changes will be made to the patient's usual anti diarrhoeal and/or anti motility agents or parenteral support during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Residual length of small bowel <200cm determined either at operation or radiologically.
* Patients with a stoma or an established enterocutaneous fistula
* Normal hydration status (urinary sodium >20mmol/L)

Exclusion Criteria:

* Dehydration (urinary sodium <20mmol/L)
* Patients with short bowel and a jejunocolonic anastomosis
* Current sepsis of any cause
* Addition/amendment to anti-diarrhoeal or anti motility agents in the last 3 days
* Severe gastrointestinal obstruction or structural abnormality of the intestine
* Active Crohn's disease - assessed using two of the three parameters:

CReactive Protein >10 Albumin <30g/L Platelets >400

* Participation in another intervention trial which may affect intestinal absorption
* Nil by mouth
* Unable or unwilling to provide consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Change in faecal sodium | Day 1 and 3
  Change in faecal sodium

CONTACTS AND LOCATIONS:
Overall Officials: alison culkin, PhD, Principal Investigator — London Northwest Healthcare Trust

IPD SHARING:
Plan to Share IPD: No